CLINICAL TRIAL: NCT05862987
Title: The Effect of Hydrogen Rich Water Intake on Acute Body Response and Following Recovery After Single 5 km Run in Endurance-untrained Men. Randomized, Double Blinded, Placebo Controlled, Cross-over Study
Brief Title: The Effect of Hydrogen Rich Water Intake on Acute Body Response and Following Recovery After 5 km Run in Untrained Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jakub Krejci, Palacky University, Faculty of Physical Culture, Palacky University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FTK_2023_14
Record Dates: First submitted 2023-05-04; First posted 2023-05-17 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Athletic Performance; Muscle Fatigue; Oxidative Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Visually indistinguishable packages of hydrogen rich water and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen rich water (Experimental): Hydrogen rich water supplied in 420 ml packages. Two days before testing - 2 packages (morning and evening), one day before testing - 3 packages (morning, afternoon, and evening), testing day - 4 packages (2 h before the run, 1 h before the run, immediately after the run, and 1 h after the run), 9 packages in total.
  Interventions: Dietary Supplement: Hydrogen rich water
- Placebo (Placebo Comparator): Tap water supplied in 420 ml packages. Two days before testing - 2 packages (morning and evening), one day before testing - 3 packages (morning, afternoon, and evening), testing day - 4 packages (2 h before the run, 1 h before the run, immediately after the run, and 1 h after the run), 9 packages in total.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrogen rich water — Hydrogen-rich water with molecular hydrogen concentration 0.9 ppm.
  Other Names: Aquastamina-R, Nutristamina, Ostrava, Czech Republic
  Arms: Hydrogen rich water
Dietary Supplement: Placebo — Tap water with molecular hydrogen concentration 0.0 ppm.
  Other Names: Aquastamina-Placebo, Nutristamina, Ostrava, Czech Republic
  Arms: Placebo

SUMMARY:
The aim of this randomized, double blinded, placebo controlled cross-over study is to evaluate the effect of hydrogen rich water intake on running performance, physiological and biochemical variables during endurance exercise and following recovery in endurance-untrained men.

DETAILED DESCRIPTION:
This study involves 16 endurance-untrained men aged 18-30 years. All participants drink hydrogen rich water (HRW) or placebo during the two days before the experiment (total volume 2100 ml) and during the testing day (total volume 1680 ml). All participants undergo one laboratory session (entry diagnostic) and two experimental sessions in the field with a washout period of 7 days. In the two experimental sessions, participants receive HRW or placebo in a randomized order. Each experimental session consisted of a pre-exercise phase, an exercise phase (5 km run), and a 24 h passive recovery phase. The following variables are assessed: running times (5 km distance and 200 m laps), heart rate, rating of perceived exertion, blood lactate, reactive strength index, subjective perceived muscle soreness, protein carbonyl content, malondialdehyde content, heart rate variability. Statistical analysis is based on analysis of variance for repeated measures with the factors water (HRW and placebo), time, and interaction. Fisher´s post hoc tests is used for pairwise comparison. The significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* No experience with endurance training.
* Good health condition.
* Signed informed content.

Exclusion Criteria:

* Acute health problems.
* Not following instructions (free of any supplements three weeks before experiment, free of any medicaments, no caffeine at least 24 hours before experiment).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Run time | Change between values before and after 7 days of crossover.
  The 5 km run is performed on a 200 m long indoor track. The running time (total time and laps times) of each runner is measured by one qualified timekeeper, which does not change between trials. The time is measured to the nearest 0.1 s with manual stopwatch.

SECONDARY OUTCOMES:
Heart rate during running | Change between values before and after 7 days of crossover.
  Heart rate during the 5 km run is continuously recorded using a heart rate monitor (Polar Team Coach, Polar, Kempele, Finland).
Rating of perceived exertion | Change between values before and after 7 days of crossover.
  The subject is asked to score subjective rating of perceived exertion using the scale developed by Borg. All subjects are familiar with the Borg scale before testing. We use the scale ranging from 6 (no exertion at all) to 20 (maximal exertion). The rating of perceived exertion is scored immediately after the run.
Blood lactate | Change between values before and after 7 days of crossover.
  Blood lactate concentration is evaluated based on blood samples taken from the fingertip. An alcohol wipe is used to clean the fingertip and the skin is punctured with a lancet. The first drop is wiped away and the second drop is used. Lactate Scout+ analyzer (EKF Diagnostics, Cardiff, United Kingdom) is used for lactate sampling. Blood lactate is evaluated after the run.
Reactive strength index | Change between values before and after 7 days of crossover.
  Reactive strength index is determined in a 5 maximum hop test performed on a mobile force platform (FP8, HUR Labs, Tampere, Finland). Each subject is instructed to maximize the jump height and minimize the ground contact time. The first hop served as a countermovement jump and is excluded from the analysis. The remaining 4 hops are averaged and reported as the outcome. The reactive strength index is determined before and after the run, 1 h and 4 h after the run.
Subjective perceived muscle soreness | Change between values before and after 7 days of crossover.
  Visual analogue scale (VAS) is used to assess lower limb muscle soreness. The VAS scale is a 100 mm long line marked with the numbers 0 (no pain) and 100 (worst imaginable pain). The VAS is assessed immediately, 1 h, 4h, and 24 h after the run.
Protein carbonyls | Change between values before and after 7 days of crossover.
  Protein carbonyls are detected from vein blood sample which is taken from the inside of the elbow by a healthcare specialist. The blood is taken into heparinized vacuum tubes. These is then centrifugated at 1000 g. Subsequently, the blood plasma is separated into cryotubes and frozen at -80 °C until biochemical analysis. Protein carbonyls concentration is determined by ELISA method in accordance with the manufacturer´s manual (Protein Carbonyl Content Assay Kit MAK094, Sigma-Aldrich, Saint Louis, USA). Protein carbonyls are sampled before and after the run, 1 h and 4 h after the run.
Malondialdehydes | Change between values before and after 7 days of crossover.
  Malondialdehydes are detected from vein blood sample which is taken from the inside of the elbow by a healthcare specialist. The blood is taken into heparinized vacuum tubes. These is then centrifugated at 1000 g. Subsequently, the blood plasma is separated into cryotubes and frozen at -80 °C until biochemical analysis. The concentration of malondialdehydes in plasma samples as lipid peroxidation products is determined using the Lipid Peroxidation Assay Kit MAK085 (Sigma-Aldrich, Saint Louis, USA) according to the manufacturer's instructions. Malondialdehydes are sampled before and after the run, 1 h and 4 h after the run.
Heart rate variability - heart rate | Change between values before and after 7 days of crossover.
  Heart rate (HR) is measured using the DiANS PF8 ECG device (DIMEA Group, Olomouc, Czech Republic). ECG sampling is performed during an orthoclinostatic maneuver in a calm room without acoustic and visual disturbances. HR is measured before and after the run, 1h and 4h after the run.
Heart rate variability - RMSSD | Change between values before and after 7 days of crossover.
  Root mean square successive difference of RR intervals (RMSSD) is measured using the DiANS PF8 ECG device (DIMEA Group, Olomouc, Czech Republic). ECG sampling is performed during an orthoclinostatic maneuver in a calm room without acoustic and visual disturbances. RMSSD is measured before and after the run, 1h and 4h after the run.
Heart rate variability - SDNN | Change between values before and after 7 days of crossover.
  Standard deviation of RR intervals (SDNN) is measured using the DiANS PF8 ECG device (DIMEA Group, Olomouc, Czech Republic). ECG sampling is performed during an orthoclinostatic maneuver in a calm room without acoustic and visual disturbances. SDNN is measured before and after the run, 1h and 4h after the run.
Heart rate variability - LF/HF | Change between values before and after 7 days of crossover.
  Ratio of low-frequency to high-frequency power (LF/HF) is measured using the DiANS PF8 ECG device (DIMEA Group, Olomouc, Czech Republic). ECG sampling is performed during an orthoclinostatic maneuver in a calm room without acoustic and visual disturbances. LF/HF is measured before and after the run, 1h and 4h after the run.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Valenta, Mgr, Principal Investigator — Palacky University
Locations (1):
- Palacky University, Faculty of Physical Culture, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw data will be made available.
Time Frame: The data will be available once the results are published in a scientific journal.
Access Criteria: For everybody.